CLINICAL TRIAL: NCT05632120
Title: Investigation of Impairments in Body Functions and Structures, Activities and Participation Restrictions According to the ICF Framework in Chronic Obstructive Pulmonary Diseases
Brief Title: Investigation of Impairments in Body Functions and Structures, Activities and Participation Restrictions in COPD
Status: Enrolling by invitation | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Istanbul Medeniyet University (Other); Biruni University (Other); Istanbul University (Other)
Responsible Party: Principal Investigator, Tansu Birinci, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: 212121
Record Dates: First submitted 2022-11-20; First posted 2022-11-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2024-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; Balance; Activity, Motor; Participation, Patient
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity; Patient Participation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This cross-sectional study aims to investigate to the impairments in body functions and structures, activities and participation restrictions according to the International Classification of Functioning, Disability and Health (ICF) framework in Chronic Obstructive Pulmonary Diseases (COPD) patients.

DETAILED DESCRIPTION:
To investigate the impairments in body functions and structures, activities and participation restrictions according to the International Classification of Functioning, Disability and Health (ICF) framework in patients with COPD, fifty patients with COPD will be included.

The Modified Medical Research Council Dyspnea (MMRC) scale and Six-Minute Walking Test (6MWT) will be used for evaluating the how dyspnea limits the patients' daily activities and functional capacity, respectively. Isometric muscle strength will be measured with a handheld dynamometer of quadriceps femoris. Fear of falling will be assessed with Activities-Specific Balance Confidence (ABC) scale. The level of dyspnea during daily activities will be assessed with London Chest Activity of Daily Living (LCADL) scale. The global impacts of COPD symptoms on overall health status will be evaluated by The COPD Assessment Test (CAT). Pulmonary function data will be retrieved from the last 1-month clinical records of the COPD patients. Statistical analysis will be performed using the Statistical Package for Social Sciences (SPSS) version 21.0. Descriptive statistics of continuous variables will be presented with mean, standard deviation (SD), confidence interval (CI) values, and descriptive statistics of categorical variables will be presented with frequency and percentage values. The conformity of the data to the normal distribution will be evaluated with the "Shapiro Wilk Test". According to the results of the analysis, "Pearson correlation test" or "Spearman correlation test" will be used to determine the relationship between dependent variables. The significance level will be set as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

1. stable disease (no severe exacerbations in the prior 3 months)
2. ability to walk independently
3. ability to read and write in Turkish
4. able to follow simple instructions
5. no pathology in visual ability and hearing

Exclusion Criteria:

1. a history of specific balance problems (i.e., diagnosed vestibular or neurological disorder)
2. severe musculoskeletal, neurological or cardiovascular disorders that limit mobility
3. use of medication(s) that may increase the risk of falls
4. participate in pulmonary rehabilitation in the lasts six months

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants will be patients with COPD diagnosed according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines were recruited from Istanbul University, Department of Chest Diseases.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Activities-Specific Balance Confidence scale | Baseline
  Activities-Specific Balance Confidence (ABC) scale will be used for evaluating the confidence in maintaining the balance in activities daily living. It provides information on the level of concern about falls during16 community-based and home-based activities. Scale scores between 0 (unsafe) to 100 (completely safe) and the total score (0-1600) is divided by 16 to obtain an individual's ABC score, with higher scores indicating greater balance confidence. In patients with COPD, the ABC scale has demonstrated construct validity as well as criterion validity for falls. In addition, the participants will be also questioned concerning the occurrence of falls and the risk of falling during the activity in each item of the ABC scale.

SECONDARY OUTCOMES:
London Chest Activity of Daily Living scale | Baseline
  London Chest Activity of Daily Living (LCADL) scale is used for assessing the level of dyspnea during daily activities.
  It is a 15-item scale comprised 4 domains: self-care (4 items), domestic (6 items), physical (2 items), and leisure (3 items). Each item scored between 0 (I wouldn't do it anyway) to 5 (I need help in doing this or someone to do it for me) and the total score ranges from 0 to 75, with higher scores indicating a more significant limitation in daily activities.
  The LCADL scale is a reliable, valid, and responsive instrument to assess limitations in performing daily activities in COPD patients. asked to rate each item in terms of risk of falling using a five-point scale, where 1=very low, 2=low, 3=moderate, 4=high, and 5=very high.
The COPD Assessment Test | Baseline
  The COPD Assessment Test (CAT) will be used for evaluating the global impacts of COPD symptoms on overall health status. Each item scores between 0 to 5 and the total score ranges from 0 to 40, with higher scores indicating the more severe impact of COPD on health status.
The strength of quadriceps femoris | Baseline
  The strength of quadriceps femoris of both sides will be measured with a hand-held dynamometer (kg.N-1) ''Nicholas Manual Muscle Tester" (model 01160, The Lafayette Instrument Company, Lafayette, Indiana). Each limb will assessed 3 times, with a recovery period of 30 seconds and the mean value will be calculated.
The Modified Medical Research Council Dyspnea scale | Baseline
  The Modified Medical Research Council Dyspnea (mMRC) scale will be used to determine how dyspnea limits the patients' daily activities performance. Itis a five-level rating scale consisting of just five items containing statements about the impact of dyspnea on the patients' daily activities performance and leading to a grade from 1 to 5. Higher scores indicate a greater impact of dyspnea on the patients' daily activities performance.
Six-Minute Walking Test (6MWT) | Baseline
  Six-Minute Walking Test (6MWT) is a reliable and valid test for evaluating functional capacity. Two 6MWTs will be performed according to the guidelines of the American Thoracic Society. The distance in meters covered over the 6 minutes of the test (6MWD) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci, PT, PhD, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University, Istanbul, Fatih/İstanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No